CLINICAL TRIAL: NCT06109753
Title: Ergonomic Benefits From Robotically Assisted Laparoscopy for Hysterectomies and Other Selected Indications in Comparison to Conventional Laparoscopy - an Explorative Study
Brief Title: Ergonomic Benefits From Robotically Assisted Laparoscopy for Hysterectomies and Other Indications
Acronym: ERCON
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Institute of Occupational and Social Medicine and Health Services Research, Tuebingen (Unknown)
Responsible Party: Sponsor
Other Study IDs: MT_ASENSUS SOS
Record Dates: First submitted 2023-10-10; First posted 2023-10-31 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Musculoskeletal Diseases or Conditions
Keywords: Muscular and mental demand; physical discomfort; eye strain
MeSH Terms: conditions — Musculoskeletal Diseases; Asthenopia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Robotically Assisted Laparoscopy: Surgeons perform robot-assisted laparoscopic surgery
  Interventions: Procedure: Robotically Assisted Laparoscopic Surgery
- Conventional Laparoscopy: Surgeons perform conventional laparoscopic surgery
  Interventions: Procedure: Conventional Laparoscopic Surgery

INTERVENTIONS:
Procedure: Robotically Assisted Laparoscopic Surgery — robotically assisted surgeries of about 60-minute duration with additional 30 min for preparing with the measurement equipment before surgery and 15 post evaluation of the corresponding surgery
  Groups: Robotically Assisted Laparoscopy
Procedure: Conventional Laparoscopic Surgery — conventional surgeries of about 60-minute duration with additional 30 min for preparing with the measurement equipment before surgery and 15 post evaluation of the corresponding surgery
  Groups: Conventional Laparoscopy

SUMMARY:
This is a prospective, single-center, observational clinical trial at the Department of Women's Health of the University Hospital Tübingen.

DETAILED DESCRIPTION:
Monocentric trial to evaluate differences in musculoskeletal and cognitive demands of robot-assisted laparoscopic surgery (RALS) vs. conventional laparoscopic surgery (CLS). Demographic and personal data are collected and pseudonymized. During surgery surface electromyography (EMG), electrocardiography (ECG), motion tracking data are collected and the surgery is documented by photos (1 photo/per second). Additionally, perceived physical discomfort (frequency and intensity) and mental load will be assessed within certain time intervals and at the very end of the surgery. The surgeon will not be disturbed in his actions and movement by the measurement equipment or applied procedures. Previous studies with similar designs can be seen as references in this context (549/2012BO1, 409/2013BO1, 262/2018BO1). After completing the surgery, the surgeon will rate difficulty of the surgery, work precision, eye strain and ergonomics during the surgery. Routine interventions like hysterectomies and other selected indications will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 68 years
* surgeons that are able to work in full shift
* trained surgeons in RALS and CLS
* written informed consent

Exclusion Criteria:

* persons influenced by analgesics or muscle relaxants
* persons not able to perform their common work for any reason
* persons with acute diseases
* muscle injury

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 4 (males and females) gynecological surgeons
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Muscle activity of the bilateral trapezius pars descendens muscle | during surgery
  The muscle activity of the bilateral trapezius pars descendens muscle will be assessed using surface electromyography, with the root-mean-square (RMS) of electrical muscle activity recordings measured through bipolar surface electrodes. Data will be normalized to an isometric voluntary maximum electrical activation (MVE).

SECONDARY OUTCOMES:
Muscle activity of the bilateral forearm muscles | during surgery
  The muscle activity of the bilateral forearm muscles will be assessed using surface electromyography, with the root-mean-square (RMS) of electrical muscle activity recordings measured through bipolar surface electrodes. Data will be normalized to an isometric voluntary maximum electrical activation (MVE).
Kinematics | during surgery
  For kinematics, the outcome measures involve the assessment of shoulder abduction, trunk, and head flexion angles in degrees, which are determined using gravimetric position sensors, providing precise measurements of body positioning during the task.
Perceived physical discomfort | during surgery
  Perceived physical discomfort is evaluated by assessing its frequency and intensity. Frequency indicates the number of occurrences, while intensity is measured on a 0 to 10 scale, where higher values indicate more intense discomfort. These measurements are recorded at 20-minute intervals to monitor changes in discomfort over time.
Perceived mental demand | during surgery
  Perceived mental demand is evaluated using the NASA (National Aeronautics and Space Administration ) Task Load Index (TLX) questionnaire's mental demand dimension, providing a subjective score ranging from 0 to 21, reflecting the perceived cognitive load during the task. Higher values are representing higher perceived mental demand.
Perceived mental demand - Heart rate | during surgery
  Heart rate (beats per minute) and heart rate variability, such as SDNN (standard deviation of the beat-to-beat differences in instantaneous heart rate), are recorded via electrocardiography to quantify physiological responses associated with mental demand.
Perceived mental demand - Heart rate variability | during surgery
  Heart rate variability, to be precise SDNN (standard deviation of the beat-to-beat differences in instantaneous heart rate), are recorded via electrocardiography to quantify physiological responses associated with mental demand.
Work precision | during surgery
  Work precision is measured during surgery using a visual analogue scale ranging from 0 to 100 mm, providing an indication of the precision and accuracy of the surgical maneuvers performed.
Eye strain | during surgery
  Eye strain is evaluated using a 10-item questionnaire designed to assess the severity of eye strain, with each question scored on a scale from 0 to 6, aiding in the comprehensive understanding of the subjective experience of visual discomfort.

OTHER OUTCOMES:
Musculoskeletal complaints | within the last 12 months
  The Nordic Questionnaire encompasses an evaluation of diverse parameters, including body height (measured in centimeters), body weight (measured in kilograms), physical activity (assessed in hours of sports per week), work experience (measured in years), and the presence of musculoskeletal complaints within the last 12 months, along with point prevalence [n]. This holistic assessment offers critical insights into the participants' physical condition and occupational health status.
  Additionally, please note that the Nordic Questionnaire does not specifically employ a single scale; rather, it utilizes various metrics tailored to the different parameters, and thus, the measurement scales can differ based on the specific parameter being assessed.
Duration of the surgical procedure | 105 Minutes
  The duration of the surgical procedure is a critical outcome measure, recorded in minutes, providing a precise indication of the time taken to complete the specific surgical intervention, aiding in the assessment of surgical efficiency and time management.
Difficulty of the surgery | 5 Minutes
  The perceived difficulty of the surgery is measured using a visual analogue scale ranging from 0 to 100 mm, with 0 indicating that the surgery was not difficult and 100 indicating that the surgery was very difficult. This measure allows the surgeons to subjectively express the complexity and challenges associated with the performed surgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Steinhilber, PD Dr., Principal Investigator — Institute of Occupational and Social Medicine and Health Services Research; Bernhard Krämer, Prof. Dr., Principal Investigator — University Women's Hospital
Locations (1):
- University Women's Hospital, Tübingen, Baden-Wurttemberg, Germany